CLINICAL TRIAL: NCT05418842
Title: Exercise Prehabilitation in Patients With Head and Neck Squamous-cell Carcinoma: The FIT4TREAT Trial
Acronym: FIT4TREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other); University Institute of Maia (Other); Aveiro University (Other); Centro Hospitalar de Vila Nova de Gaia/Espinho (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F4T
Record Dates: First submitted 2022-05-16; First posted 2022-06-14 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Neoplasms
Keywords: Prehabilitation; Exercise; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Group (Experimental): In addition to standard medical care, the prehabilitation group will have three supervised exercise training sessions per week from diagnosis to start of radiotherapy (pre-treatment phase).
  Interventions: Other: Prehabilitation
- Control Group (No Intervention): The control group will receive the standard medical care.

INTERVENTIONS:
Other: Prehabilitation — In addition to usual care, the prehabilitation group will exercise 3 times a week, starting immediately after diagnosis and throughout the pre-treatment period. Each exercise session will encompass 5-min warm-up and 45-min conditioning exercises. Aerobic training will be performed using low-volume high intensity interval training (HIIT). The HIIT duration is 16-20 minutes and it will be performed with 8-10 intervals of high intensity (1 minute) and 8-10 intervals of low intensity (1 minute). High intensity intervals will be set to an external load that represents 85-90% of estimated VO2Peak. In addition, patients will do resistance training at moderate intensity. Patients will complete 2 sets of 12 repetitions of 5 upper and lower body exercises.
  Arms: Prehabilitation Group

SUMMARY:
The main purpose of this randomized-controlled trial is to evaluate the effects of prehabilitation based on exercise training (ET) on functional capacity in HNC patients treated with chemoradiotherapy (CRT). Forty-six participants will be randomized (1:1 ratio) into prehabilitation and usual care groups. The length of intervention will be at least 2 weeks. Data will be collected at diagnosis, immediately before anti-cancer treatment start and 4 weeks following CRT. Primary outcome is functional capacity as assessed by the six-minute walk test. Additional measures include muscle strength, endothelial function, arterial stiffness, inflammatory biomarkers, body composition, quality of life, treatment tolerance, compliance to treatment, progression-free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Histologically confirmed HNSCC located on the oral cavity, larynx, oropharynx, hypopharynx, nasopharynx or in lymph nodes from an unknown primary tumor (stage I-IV);
* Proposed for concomitant chemoradiotherapy with curative intent;
* Date of treatment beginning ≥2 weeks from baseline assessment;
* ECOG-Performance Status 0-1.

Exclusion Criteria:

* Completion of previous anticancer treatment within less than a year;
* Uncontrolled hypertension, cardiac or pulmonary disease;
* Contraindications to exercise training;
* Inability to provide informed consent;
* Expected inability to fulfil the proposed schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by six-minute walk test.

SECONDARY OUTCOMES:
Functional Capacity | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by six-minute walk test.
Isometric Handgrip Muscle Strength | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by hand dynamometer.
Isometric Handgrip Muscle Strength | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by hand dynamometer.
Arterial Stiffness | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by carotid-femoral pulse wave velocity.
Arterial Stiffness | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by carotid-femoral pulse wave velocity.
Endothelial Function | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by brachial artery dilation to endothelial-dependent stimuli using an ultrasound, according to the recommendations.
Endothelial Function | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by brachial artery dilation to endothelial-dependent stimuli using an ultrasound, according to the recommendations.
Lower Limb Functionality | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by 30-second sit to stand test.
Lower Limb Functionality | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by 30-second sit to stand test.
Health-related Quality of Life | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include 5 functional scales, 3 symptom scales, a global health status / QoL scale, and 6 single items. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Health-related Quality of Life | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include 5 functional scales, 3 symptom scales, a global health status / QoL scale, and 6 single items. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Head and Neck Cancer-specific Quality of Life | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN43). This is the head and neck cancer specific module that contains 43 questions with 19 symptoms scales. All of the multi-item scales and single-item measures range in score from 0 to 100. A high score represents a high level of symptomatology or problems.
Head and Neck Cancer-specific Quality of Life | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN43). This is the head and neck cancer specific module that contains 43 questions with 19 symptoms scales. All of the multi-item scales and single-item measures range in score from 0 to 100. A high score represents a high level of symptomatology or problems.
Body Weight | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by bioelectrical impedance.
Body Weight | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by bioelectrical impedance.
Body Mass Index | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by participant's weight in kilograms divided by the square of height in meters.
Body Mass Index | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by participant's weight in kilograms divided by the square of height in meters.
Muscle Mass | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by bioelectrical impedance.
Muscle Mass | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by bioelectrical impedance.
Percentage of Body Fat | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
  Assessed by bioelectrical impedance.
Percentage of Body Fat | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
  Assessed by bioelectrical impedance.
C-Reactive Protein | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
C-Reactive Protein | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
Albumin | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
Albumin | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
Hemogram | Change from Baseline (at diagnosis) to 1-3 days before the beginning of radiotherapy
Hemogram | Change from 1-3 days before the beginning of radiotherapy to 4 Weeks after last radiotherapy session
Unplanned hospital visits | From baseline to 4 Weeks after last radiotherapy session
Compliance to Chemotherapy | Through chemotherapy completion, an average of 7 weeks
  Assessed as the average relative chemotherapy dose-intensity received for the originally planned regimen based on standard formulas.
Compliance to Radiotherapy | Through radiotherapy completion, an average of 7 weeks
  Assessed assessed as the completion of prescribed dose of radiation during the prescribed time frame.
Treatment-Related Adverse Events | From the beginning of radiotherapy/chemotherapy to 4 Weeks after last radiotherapy session
  Assessed by CTCAE-vs.5.
Progression-Free Survival | From baseline to 5 years after diagnosis
  Defined as the time from randomization to the occurrence of disease progression or death.
Overall Survival | From baseline to 5 years after diagnosis
  Defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Garcia, Msc, Principal Investigator — Research Center of Sports Science Health Science and Human Development - University of Maia
Locations (5):
- Portugal (5):
  - University of Maia, Maia, Porto District
  - Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Porto District
  - Instituto Português de Oncologia do Porto (IPO-Porto), Porto, Região
  - University of Aveiro, Aveiro
  - Liga Portuguesa Contra o Cancro - Núcleo Regional do Norte (LPCC-NRN), Porto